CLINICAL TRIAL: NCT01837797
Title: Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose Study to Evaluate the Efficacy and Safety of Brexpiprazole (1 and 3 mg/Day) as Adjunctive Treatment in Elderly Patients With Major Depressive Disorder With an Inadequate Response to Antidepressant Treatment
Brief Title: Efficacy and Safety of Brexpiprazole as Adjunctive Treatment in Elderly Patients With Major Depressive Disorder With an Inadequate Response to Antidepressant Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated because of recruitment challenges
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14571A; 2012-001361-32 (EudraCT Number)
Record Dates: First submitted 2013-04-04; First posted 2013-04-23 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Interventions: Drug: Placebo
- Brexpiprazole 1 mg (Experimental): Brexpiprazole adjunct to open-label treatment with a commercially available ADT. Brexpiprazole dosing was 0.5 mg/day in the first 1 week followed by 1 mg/day.
  Interventions: Drug: Brexpiprazole 1 mg
- Brexpiprazole 3 mg (Experimental): Brexpiprazole adjunct to open-label treatment with a commercially available ADT. Brexpiprazole dosing was 0.5 mg/day in the first 1 week, 1 mg/day in the second week, followed by 3 mg/day.
  Interventions: Drug: Brexpiprazole 3 mg

INTERVENTIONS:
Drug: Placebo — Once daily, tablets, orally
  Arms: Placebo
Drug: Brexpiprazole 1 mg — once daily dose, tablets, orally
  Arms: Brexpiprazole 1 mg
Drug: Brexpiprazole 3 mg — once daily dose, tablets, orally
  Arms: Brexpiprazole 3 mg

SUMMARY:
To evaluate the efficacy and safety of brexpiprazole as adjunctive treatment in elderly patients with Major Depressive Disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* The patient is an outpatient consulting a psychiatrist.
* The patient has a recurrent Major Depressive Disorder diagnosed according to DSM-IV-TR™. The current Major Depressive Episode (MDE) should be confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient had at least one previous MDE before the age of 60 years.
* The patient has a moderate to severe depression and an insufficient response to at least one and no more than three adequate antidepressants treatments.
* The patient, if a woman, must have had her last natural menstruation ≥24 months prior to the Screening Visit.
* The patient, if a man, agrees to protocol-defined use of effective contraception if his female partner is of childbearing potential.

Exclusion Criteria:

* The patient has any current psychiatric disorder or Axis I disorder (DSM-IV-TR™ criteria), established as the primary diagnosis, other than MDD.
* The patient has a current Axis II (DSM-IV-TR™) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypical or histrionic personality disorder.
* The patient has experienced/experiences hallucinations, delusions or any psychotic symptomatology in the current MDE.
* The patient suffers from mental retardation, organic mental disorders, or mental disorders due to a general medical condition (DSM-IV-TR™ criteria).
* The patient, in the opinion of the investigator, or according to Columbia Suicide Severity Rating Scale (C-SSRS), is at significant risk of suicide.
* The patient has had neuroleptic malignant syndrome.
* The patient has any relevant medical history or current presence of systemic disease.
* The patient has a neurodegenerative disorder.
* The patient has, at the Screening Visit an abnormal ECG that is, in the investigator's opinion, clinically significant.
* The patient has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin, that has not been in remission for >5 years prior to the first dose of IMP.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (2):
- United States (2):
  - US001, National City, California
  - US008, Orlando, Florida

REFERENCES:
- See also: EMA EudraCT Result Posting — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-001361-32/results

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 129 patients were enrolled in the study and 128 patients received open-label treatment with one of six commercially available antidepressant antidepressant treatments (ADT) together with double-blind study treatment. Only 15 patients were randomized to Period 2 before the study was terminated; 47 patients entered Period 3.
Groups:
- Period 1 Placebo and ADT; Period 2 Placebo and ADT: Placebo adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Placebo: Once daily, tablets, orally
- Period 2 Brexpiprazole 1 mg and ADT: Brexpiprazole 1 mg adjunct to open-label treatment with a commercially available ADT
  Brexpiprazole: 1 mg once daily, tablets, orally
- Period 2 Brexpiprazole 3 mg and ADT: Brexpiprazole 3 mg adjunct to open-label treatment with a commercially available ADT
  Brexpiprazole: 3 mg once daily, tablets, orally
- Period 3 Placebo and ADT: Placebo adjunct to open-label treatment with commercially available antidepressant treatment (ADT)
  Placebo: Once daily, tablets, orally
Period: Period 1
Arm/Group | Period 1 Placebo and ADT | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT | Period 3 Placebo and ADT
Started | 129 | 0 | 0 | 0 | 0
Completed | 27 | 0 | 0 | 0 | 0
Not Completed | 102 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 0 | 0
Not completed — Administrative reasons | 76 | 0 | 0 | 0 | 0
Not completed — Withdrawal of consent before treatment | 1 | 0 | 0 | 0 | 0
Not completed — Other | 10 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Period 1 Placebo and ADT | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT | Period 3 Placebo and ADT
Started | 0 | 6 | 3 | 6 | 0
Completed | 0 | 1 | 1 | 1 | 0
Not Completed | 0 | 5 | 2 | 5 | 0
Not completed — Administrative or other reasons | 0 | 5 | 2 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Period 1 Placebo and ADT | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT | Period 3 Placebo and ADT
Started | 0 | 0 | 0 | 0 | 47
Completed | 0 | 0 | 0 | 0 | 24
Not Completed | 0 | 0 | 0 | 0 | 23
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Administrative reasons | 0 | 0 | 0 | 0 | 20
Not completed — Other | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Period 2 Brexpiprazole 1 mg and ADT: Brexpiprazole 1 mg adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Brexpiprazole: 1 mg once daily, tablets, orally
- Period 2 Brexpiprazole 3 mg and ADT: Brexpiprazole 3 mg adjunct to open-label treatment with a commercially available antidepressant (ADT)
  Brexpiprazole: 3 mg once daily, tablets, orally
- Total: Total of all reporting groups
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT | Total
Number analyzed (Participants) | 6 | 3 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 6 | 3 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 6 | 11
  Male | 3 | 1 | 0 | 4

OUTCOME MEASURES:

1. Secondary Outcome: Number of Adverse Events
Description: 15 patients were enrolled to Period 2; only 3 patients completed due to study termination
Time Frame: From randomisation to follow-up (week 24)
Measure: Number; unit: Adverse events
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 6 | 3 | 6
Adverse events | 3 | 5 | 2

2. Primary Outcome: Change From Randomisation in Depressive Symptoms During the Randomised Treatment
Description: Montgomery and Aasberg Depression Rating Scale (MADRS) total score
Time Frame: From randomisation to end of treatment (week 20)
Population: Only 3 patients completed study Period 2. A total of 129 patients were enrolled when the study was terminated (Planned: 1334 patients). The limited number of enrolled patients would result in insufficient data for analyses, therefore, no data were collected
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Randomisation in Clinical Global Impression During the Randomised Treatment
Description: Clinical Global Impression - Severity of illness (CGI-S) score
Time Frame: From randomisation to end of treatment (week 20)
Population: as for outcome 2
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Randomisation in Functionality Assessed by SDS During the Randomised Treatment
Description: Sheehan Disability Scale (SDS) total score
Time Frame: From randomisation to end of treatment (week 20)
Population: as for outcome 2
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Randomisation in Social Adaptation During the Randomised Treatment
Description: Social Adaptation Self-evaluation Scale (SASS) total score
Time Frame: From randomisation to end of treatment (week 20)
Population: as for outcome 2
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Response During the Randomised Treatment
Description: Based on a pre-specified decrease in MADRS total score
Time Frame: From randomisation to end of treatment (week 20)
Population: as for outcome 2
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Sustained Response During the Randomised Treatment
Description: Based on a pre-specified decrease in MADRS total score
Time Frame: From randomisation to end of treatment (week 20)
Population: as for outcome 2
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Remission During the Randomised Treatment
Description: Based on a pre-specified MADRS total score
Time Frame: From randomisation to end of treatment (week 20)
Population: as for outcome 2
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Sustained Remission During the Randomised Treatment
Description: Based on a pre-specified MADRS total score
Time Frame: From randomisation to end of treatment (week 20)
Population: as for outcome 2
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Patients With Risk of Suicidality Assessed Using the Electronic Columbia Suicide Severity Rating Scale (eC-SSRS)
Description: The Columbia Suicide Severity Rating Scale (eC-SSRS) is a semi-structured interview developed to systematically assess suicidal ideation and behaviour of patients participating in a clinical study. The C-SSRS has 5 questions addressing suicidal ideation, 5 sub-questions assessing the intensity of ideation, and 4 questions addressing suicidal behaviour.
Time Frame: From randomisation to end of treatment (week 20)
Population: 15 patients were enrolled to Period 2, only 3 patients completed due to study termination
Measure: Number; unit: participants
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Number analyzed (Participants) | 6 | 3 | 6
participants
  No suicidal ideation or behaviour | 6 | 3 | 4
  Any non-suicidal self-injurious behavior | 0 | 0 | 0
  Suicidal Ideation | 0 | 0 | 2
  Preparatory action towards imminent suicidal behav | 0 | 0 | 0
  Not fatal suicide attempt | 0 | 0 | 0
  Completed suicide | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization to follow-up
Arm/Group | Period 2 Placebo and ADT | Period 2 Brexpiprazole 1 mg and ADT | Period 2 Brexpiprazole 3 mg and ADT
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 2/3 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 2 Placebo and ADT (N=6) | Period 2 Brexpiprazole 1 mg and ADT (N=3) | Period 2 Brexpiprazole 3 mg and ADT (N=6)
Gait disturbance (General disorders) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Bruxism (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Because the study was terminated, few efficacy data were collected. These data have not been reported in accordance with the ICH E3 regarding abbreviated clinical study reports. Furthermore, no firm conclusions can be drawn regarding safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No